CLINICAL TRIAL: NCT01349361
Title: Treatment of Basal Cell Carcinomas With Methyl Aminolevulinate and Daylight
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Hans Christian Wulf, Bispebjerg Hospital
Other Study IDs: 2010-024517-31
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-03

CONDITIONS: Photodynamic Therapy; Basal Cell Carcinomas
MeSH Terms: conditions — Carcinoma, Basal Cell

ARMS (1):
- Daylight-PDT (Experimental)
  Interventions: Procedure: Daylight mediated photodynamic therapy

INTERVENTIONS:
Procedure: Daylight mediated photodynamic therapy

SUMMARY:
Photodynamic Therapy (PDT) is an effective treatment of basal cell carcinomas (BCC) however the inconvenience of clinic attendance and discomfort during therapy are significant drawbacks. The objective of this study is to evaluate the effect of daylight-mediated PDT of BCC.

ELIGIBILITY:
Inclusion Criteria:

* superficial BCC

Exclusion Criteria:

* Immunosuppression

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2011-03; Primary Completion 2013-01

PRIMARY OUTCOMES:
complete disappearance of the BCC

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark